CLINICAL TRIAL: NCT04546789
Title: Phase I Open-label, Single Dose Study to Investigate the Effect of Hepatic Impairment on the PK of Evobrutinib (M2951)
Brief Title: Effect of Hepatic Impairment on M2951 (BTK Inhibitor) PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS200527_0059; 2020-001920-32 (EudraCT Number)
Record Dates: First submitted 2020-09-10; First posted 2020-09-14 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Pharmacokinetics
MeSH Terms: interventions — evobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Normal Hepatic Function (Reference) (Experimental): Participants with normal hepatic function received single oral dose of 30 milligrams (mg) M2951 (3 film-coated tablets of 10 mg) on Day 1 after a standard breakfast.
  Interventions: Drug: M2951 (BTK inhibitor)
- Group 2: Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment (Child-Pugh Class A, score 5 to 6) received single oral dose of 30 mg M2951 (3 film-coated tablets of 10 mg) on Day 1 after a standard breakfast. The Child-Pugh Score was a scoring system used to determine the prognosis with cirrhosis and need for liver transplantation. Scoring is based upon serum albumin, ascites, serum bilirubin, prothrombin time, and encephalopathy. Each category is based on a scoring system of 1-3 with 3 being the worst and a total score range of 5-15. It is broken into categories A (score of 5-6), B (score of 7-9), and C (score of 10-15) with worsening from A to C for prognosis.
  Interventions: Drug: M2951 (BTK inhibitor)
- Group 3: Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (Child-Pugh Class B, score 7 to 9) received single oral dose of 30 mg M2951 (3 film-coated tablets of 10 mg) on Day 1 after a standard breakfast. The Child-Pugh Score was a scoring system used to determine the prognosis with cirrhosis and need for liver transplantation. Scoring is based upon serum albumin, ascites, serum bilirubin, prothrombin time, and encephalopathy. Each category is based on a scoring system of 1-3 with 3 being the worst and a total score range of 5-15. It is broken into categories A (score of 5-6), B (score of 7-9), and C (score of 10-15) with worsening from A to C for prognosis.
  Interventions: Drug: M2951 (BTK inhibitor)

INTERVENTIONS:
Drug: M2951 (BTK inhibitor) — Participants received a single oral dose of M2951 (BTK inhibitor) on Day 1.
  Other Names: Evobrutinib

SUMMARY:
This study was to investigate the pharmacokinetic (PK) and safety of M2951 (Bruton's tyrosine kinase [BTK] inhibitor) in participants with different degrees of hepatic impairment compared to participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Participants with normal hepatic function only will be overtly healthy as determined by medical evaluation, including no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion OR
* Participants with moderately impaired hepatic function only will be considered to have moderately (Child-Pugh class B and confirmed liver cirrhosis) impaired hepatic function and has been clinically stable for at least 1 month prior to Screening OR
* Participants with mildly impaired hepatic function only will be considered to have mildly (Child-Pugh class A and confirmed liver cirrhosis) impaired hepatic function and has been clinically stable for at least 1 month prior to Screening
* Have a body weight within 50.0 and 120.0 kilogram (kg) and body mass index (BMI) within the range 19.0 and 36.0 kilogram per square meter (kg/m^2)
* Female participants are not pregnant or breastfeeding, and at least one of the following conditions applies
* Not a woman of childbearing potential (WOCBP)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Clinical history of autoimmune disorder with hepatic influence (Hashimoto thyroiditis and rheumatic diseases allowed)
* History of any malignancy
* Diseases and surgeries of the gastrointestinal tract, which could influence the gastrointestinal anatomy and mobility. Prior history of cholecystectomy or inflammatory bowel disease, and any clinically relevant surgery within 6 months prior to Screening
* History of chronic or recurrent acute infection or any bacterial, viral, parasitic or fungal infections within 30 days prior to Screening and at any time between Screening and admission, or hospitalization due to infection within 6 months prior to Screening
* History of shingles within 12 months prior to Screening
* History of drug hypersensitivity, ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients; history of serious allergic reactions leading to hospitalization or any other hypersensitivity reaction in general, which may affect the safety of the participant and/or outcome of the trial per the Investigator's discretion
* Participants with impaired hepatic function will be excluded who had Primary and secondary biliary cirrhosis.
* Participants with impaired hepatic function will be excluded with Clinical evidence of severe ascites.
* Participants with impaired hepatic function will be excluded with Hepatic encephalopathy Grade greater than 1
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2021-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0059
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 32 participants were screened. Out of which, 24 participants were enrolled and treated in the study.
Groups:
- Group 2: Mild Hepatic Impairment (Child-Pugh Class A): Participants with mild hepatic impairment (Child-Pugh Class A, score 5 to 6) received single oral dose of 30 mg M2951 (3 film-coated tablets of 10 mg) on Day 1 after a standard breakfast. The Child-Pugh Score was a scoring system used to determine the prognosis with cirrhosis and need for liver transplantation. Scoring is based upon serum albumin, ascites, serum bilirubin, prothrombin time, and encephalopathy. Each category is based on a scoring system of 1-3 with 3 being the worst and a total score range of 5-15. It is broken into categories A (score of 5-6), B (score of 7-9), and C (score of 10-15) with worsening from A to C for prognosis.
- Group 3: Moderate Hepatic Impairment (Child-Pugh Class B): Participants with moderate hepatic impairment (Child-Pugh Class B, score 7 to 9) received single oral dose of 30 mg M2951 (3 film-coated tablets of 10 mg) on Day 1 after a standard breakfast. The Child-Pugh Score was a scoring system used to determine the prognosis with cirrhosis and need for liver transplantation. Scoring is based upon serum albumin, ascites, serum bilirubin, prothrombin time, and encephalopathy. Each category is based on a scoring system of 1-3 with 3 being the worst and a total score range of 5-15. It is broken into categories A (score of 5-6), B (score of 7-9), and C (score of 10-15) with worsening from A to C for prognosis.
Period: Overall Study
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis population (SAF) included all participants who were administered any dose of any study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (5.70) | 58.4 (11.30) | 58.9 (10.40) | 60.8 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 5 | 4 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 8 | 8 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of M2951
Description: AUC0-inf was calculated by combining AUC0-tlast and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 32.0 hours post-dose
Population: The Pharmacokinetic Analysis Population (PK) was a subset of the SAF analysis population and consisted of all participants who received at least one dose of active Investigational Medicinal Product (IMP) and provide at least one measurable post-dose concentration. A measurement below lower limit of quantification (BLQ) is considered a valid measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
hour*nanogram per milliliter (h*ng/mL) | 186 (23.6) | 232 (60.6) | 362 (21.8)
Statistical Analysis 1: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 2: Mild Hepatic Impairment (Child-Pugh Class A); Mild Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least squares mean = 1.25, 90% CI 2-sided [0.86 to 1.82]
Statistical Analysis 2: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 3: Moderate Hepatic Impairment (Child-Pugh Class B); Moderate hepatic impairment vs Normal hepatic impairment; Test type: Other; Ratio of geometric least square mean = 1.95, 90% CI 2-sided [1.60 to 2.38]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of M2951
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 32.0 hours post-dose
Population: The PK population was a subset of the SAF analysis population and consisted of all participants who received at least one dose of active IMP and provide at least one measurable post-dose concentration. A measurement BLOQ is considered a valid measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
nanogram per milliliter (ng/mL) | 63.8 (14.2) | 79.2 (86.2) | 118 (29.9)
Statistical Analysis 1: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 2: Mild Hepatic Impairment (Child-Pugh Class A); Mild Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 1.24, 90% CI 2-sided [0.77 to 1.99]
Statistical Analysis 2: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 3: Moderate Hepatic Impairment (Child-Pugh Class B); Moderate Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 1.85, 90% CI 2-sided [1.51 to 2.26]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as events that started or worsened that in severity after at least one dose of the study intervention has been administered. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: up to follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 1

4. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets and Reticulocytes
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the hematology parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils, platelets and reticulocytes. Change from baseline in hematology parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils, platelets, and reticulocytes at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
10^9 cells per liter
  Basophils: Day 2 | -0.006 (0.0160) | -0.005 (0.0107) | -0.003 (0.0175)
  Basophils: follow- up (Day 6) | -0.003 (0.0128) | 0.004 (0.0119) | 0.006 (0.0119)
  Eosinophils: Day 2 | -0.007 (0.0984) | -0.025 (0.0568) | 0.010 (0.0650)
  Eosinophils: follow- up (Day 6) | 0.000 (0.0626) | -0.040 (0.0518) | 0.016 (0.1051)
  Leukocytes: Day 2 | 0.54 (0.597) | -0.28 (0.504) | -0.68 (1.074)
  Leukocytes: follow- up (Day 6) | 0.11 (0.751) | -0.10 (0.857) | -0.66 (1.265)
  Lymphocytes: Day 2 | 0.233 (0.3186) | -0.055 (0.1099) | 0.141 (0.3541)
  Lymphocytes: follow- up (Day 6) | 0.146 (0.3074) | 0.046 (0.1994) | 0.024 (0.2900)
  Monocytes: Day 2 | 0.004 (0.0752) | 0.009 (0.0930) | -0.076 (0.1905)
  Monocytes: follow- up (Day 6) | 0.008 (0.0761) | 0.071 (0.1173) | -0.033 (0.1618)
  Neutrophils: Day 2 | 0.300 (0.4459) | -0.186 (0.4348) | -0.744 (0.9999)
  Neutrophils: follow- up (Day 6) | -0.043 (0.8141) | -0.169 (0.7111) | -0.659 (1.1235)
  Platelets: Day 2 | -3.3 (21.12) | -16.5 (13.72) | -27.3 (18.73)
  Platelets: follow- up (Day 6) | -7.0 (21.85) | -12.0 (9.80) | -22.3 (23.89)
  Reticulocytes: Day 2 | 3.50 (5.025) | -1.97 (9.358) | -5.01 (7.052)
  Reticulocytes: follow- up (Day 6) | 2.51 (7.248) | -3.14 (4.541) | 4.76 (10.136)

5. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes, Neutrophils/Leukocytes and Reticulocytes/Erythrocytes
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the hematology parameters: basophils/leukocytes, eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes, neutrophils/leukocytes and reticulocytes/erythrocytes. Change From Baseline in hematology parameters: basophils/leukocytes, eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes, neutrophils/leukocytes and reticulocytes/erythrocytes at Day 2 and Day 6 were reported in percentage.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
percentage of cells
  Basophils/Leukocytes: Day 2 | -0.16 (0.185) | -0.04 (0.207) | 0.01 (0.323)
  Basophils/Leukocytes: follow- up (Day 6) | -0.08 (0.212) | 0.06 (0.283) | 0.21 (0.348)
  Eosinophils/Leukocytes: Day 2 | -0.33 (1.285) | -0.29 (0.933) | 0.31 (1.249)
  Eosinophils/Leukocytes: follow- up (Day 6) | -0.04 (0.924) | -0.45 (0.802) | 0.50 (1.379)
  Lymphocytes/Leukocytes: Day 2 | 0.95 (3.575) | -0.18 (1.689) | 3.66 (6.029)
  Lymphocytes/Leukocytes: follow- up (Day 6) | 1.49 (6.414) | 1.25 (2.968) | 2.26 (4.562)
  Monocytes/Leukocytes: Day 2 | -0.59 (1.034) | 0.39 (1.578) | 0.04 (1.550)
  Monocytes/Leukocytes: follow- up (Day 6) | -0.11 (0.989) | 1.33 (1.433) | 0.56 (2.042)
  Neutrophils/Leukocytes: Day 2 | 0.12 (4.556) | 0.11 (3.328) | -4.02 (6.968)
  Neutrophils/Leukocytes: follow- up (Day 6) | -1.26 (7.166) | -2.19 (4.008) | -3.54 (7.499)
  Reticulocytes/Erythrocyte: Day 2 | 0.076 (0.1131) | 0.008 (0.1978) | -0.083 (0.1581)
  Reticulocytes/Erythrocyte: follow- up (Day 6) | 0.085 (0.1640) | 0.006 (0.1314) | 0.210 (0.3447)

6. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Change from baseline in hematology parameter: erythrocytes mean corpuscular hemoglobin at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
picogram
  Day 2 | -0.04 (0.307) | -0.25 (0.389) | -0.07 (0.373)
  Follow- up (Day 6) | -0.09 (0.348) | -0.02 (0.225) | 0.06 (0.487)

7. Secondary Outcome: Change From Baseline in Hematology Parameters: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the hematology parameter: erythrocytes mean corpuscular volume. Change from baseline in hematology parameter: erythrocytes mean corpuscular volume at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
femtoliters
  Day 2 | 0.14 (0.983) | 0.03 (1.562) | -0.22 (1.445)
  Follow- up (Day 6) | 0.61 (0.969) | 0.54 (0.940) | -0.19 (0.662)

8. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the hematology parameters: erythrocytes. Change from baseline in hematology parameters: erythrocytes at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
10^12 cells per liter
  Day 2 | 0.017 (0.1945) | -0.096 (0.2894) | -0.113 (0.2858)
  Follow- up (Day 6) | -0.083 (0.1348) | -0.163 (0.1992) | -0.179 (0.1787)

9. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the hematology parameter: hematocrit. Change from baseline in hematology parameter: hematocrit at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: liter of cells per liter of blood (L/L)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
liter of cells per liter of blood (L/L)
  Day 2 | 0.0022 (0.01795) | -0.0096 (0.02650) | -0.0112 (0.03179)
  Follow- up (Day 6) | -0.0042 (0.01059) | -0.0131 (0.01840) | -0.0174 (0.01683)

10. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the hematology parameter: hemoglobin. Change from baseline in hematology parameter: hemoglobin at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
gram per liter (g/L)
  Day 2 | 0.4 (5.55) | -4.5 (10.43) | -3.6 (9.23)
  Follow- up (Day 6) | -2.9 (3.94) | -5.6 (6.82) | -5.4 (4.44)

11. Secondary Outcome: Change From Baseline in Hematology Parameter: Prothrombin International Normalized Ratio
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the hematology parameter: Prothrombin International Normalized Ratio. International Normalized Ratio (INR) is calculated based on the prothrombin time (PT) test results. The INR is the ratio of a participant's prothrombin time to a normal (control) sample, raised to the power of the International Sensitivity Index (ISI) value for the analytical system being used. Change from baseline in hematology parameter: prothrombin international normalized ratio at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
ratio
  Day 2 | -0.006 (0.0160) | 0.006 (0.0262) | 0.006 (0.0421)
  Follow- up (Day 6) | 0.021 (0.0295) | -0.006 (0.0580) | -0.029 (0.0391)

12. Secondary Outcome: Change From Baseline in Hematology Parameter: Prothrombin Time
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the hematology parameter: prothrombin time. Prothrombin Time measures how long it takes for a clot to form in a blood sample. Change from baseline in hematology parameter: prothrombin time at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
seconds
  Day 2 | -0.12 (0.183) | 0.04 (0.245) | 0.14 (0.396)
  Follow- up (Day 6) | 0.12 (0.337) | -0.06 (0.510) | -0.19 (0.336)

13. Secondary Outcome: Change From Baseline in Chemistry Parameters: Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Aspartate Aminotransferase, Creatine Kinase, Gamma Glutamyl Transferase, Lactate Dehydrogenase, Lipase
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the chemistry parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Amylase, Aspartate Aminotransferase (AST), Creatine Kinase (CK), Gamma Glutamyl Transferase (GGT), Lactate Dehydrogenase (LDH) and Lipase. Change from baseline in chemistry parameters: ALT, ALP, Amylase, AST, CK, GGT, LDH and Lipase at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: units per litre (U/L)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
units per litre (U/L)
  ALT: Day 2 | 0.9 (2.23) | -9.4 (17.00) | -2.0 (3.82)
  ALT: follow- up (Day 6) | 0.8 (2.12) | -7.0 (20.50) | -0.4 (2.13)
  ALP: Day 2 | -3.3 (5.47) | -14.6 (16.04) | -16.1 (13.17)
  ALP: follow- up (Day 6) | 0.4 (5.66) | -9.5 (14.06) | -9.5 (19.27)
  Amylase: Day 2 | 1.8 (15.71) | -11.0 (8.32) | 34.1 (107.34)
  Amylase: follow- up (Day 6) | -4.1 (6.47) | -2.6 (3.46) | 14.1 (21.56)
  AST: Day 2 | -0.5 (2.88) | -24.1 (51.88) | 2.1 (7.38)
  AST: follow- up (Day 6) | 0.6 (1.92) | -15.5 (51.39) | 0.8 (5.01)
  CK: Day 2 | -41.9 (40.65) | -68.0 (27.44) | -36.4 (23.08)
  CK: follow- up (Day 6) | -20.9 (44.97) | -15.4 (26.42) | -9.5 (43.36)
  GGT: Day 2 | -0.8 (1.39) | -22.4 (34.98) | 6.5 (52.11)
  GGT: follow- up (Day 6) | -1.0 (1.85) | -24.8 (43.48) | -27.6 (43.00)
  LDH: Day 2 | -17.6 (17.44) | -42.5 (35.62) | -11.3 (33.72)
  LDH: follow- up (Day 6) | -13.9 (10.44) | -20.9 (23.73) | -10.8 (12.71)
  Lipase: Day 2 | 18.4 (50.86) | -4.8 (3.62) | -16.8 (63.92)
  Lipase: follow- up (Day 6) | -2.4 (7.05) | -1.5 (5.35) | 10.4 (28.61)

14. Secondary Outcome: Change From Baseline in Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the chemistry parameters: Albumin and Protein. Change from baseline in chemistry parameters: albumin and protein level at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
g/L
  Albumin: Day 2 | -1.1 (2.64) | -4.0 (3.74) | -2.3 (3.11)
  Albumin: follow- up (Day 6) | -0.6 (2.00) | -1.5 (2.73) | -0.8 (0.89)
  Protein: Day 2 | -1.3 (3.11) | -6.0 (5.98) | -3.3 (4.86)
  Protein: follow- up (Day 6) | -1.0 (2.88) | -2.8 (4.92) | -1.5 (1.93)

15. Secondary Outcome: Change From Baseline in Chemistry Parameters: Bilirubin, Creatinine and Urate
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the chemistry parameters: Bilirubin, Creatinine and Urate. Change from baseline in chemistry parameters: bilirubin, creatinine and urate level at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
micromole per liter (mcmol/L)
  Bilirubin: Day 2 | -0.42760 (1.516108) | 3.41455 (7.539097) | 3.20700 (7.993130)
  Bilirubin: follow- up (Day 6) | 0.21380 (2.131883) | -0.21380 (5.593931) | -2.77940 (6.060122)
  Creatinine: Day 2 | -7.0720 (5.21913) | -3.0940 (5.88280) | -5.3040 (5.78714)
  Creatinine: follow- up (Day 6) | -0.0000 (4.84187) | 1.7680 (4.77220) | -0.4420 (2.87421)
  Urate: Day 2 | -25.2790 (28.03413) | -24.5355 (35.89100) | -15.6135 (28.06792)
  Urate: follow- up (Day 6) | 5.9480 (38.80879) | -11.8960 (25.82908) | 8.9220 (18.80923)

16. Secondary Outcome: Change From Baseline in Chemistry Parameter: C Reactive Protein
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the chemistry parameter: C Reactive Protein. Change from baseline in chemistry parameters: C Reactive Protein level at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
milligram per liter (mg/L)
  Day 2 | -0.04 (0.460) | -0.22 (0.669) | 0.40 (1.593)
  Follow- up (Day 6) | -0.05 (0.404) | 0.26 (0.798) | 1.25 (2.330)

17. Secondary Outcome: Change From Baseline in Chemistry Parameters: Calcium, Chloride, Cholesterol, Glucose, Magnesium, Phosphate, Potassium, Sodium, Triglycerides, Urea and Urea Nitrogen
Description: Blood samples were collected in a fasted condition (after a fast of at least 8 hours) to analyze the chemistry parameters: Calcium, Chloride, Cholesterol, Glucose, Magnesium, Phosphate, Potassium, Sodium, Triglycerides, Urea and Urea Nitrogen. Change from baseline in chemistry parameters: Calcium, Chloride, Cholesterol, Glucose, Magnesium, Phosphate, Potassium, Sodium, Triglycerides, Urea and Urea Nitrogen level at Day 2 and Day 6 were reported.
Time Frame: Baseline, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
millimole per liter (mmol/L)
  Calcium: Day 2 | -0.030 (0.0481) | -0.020 (0.0878) | -0.036 (0.0540)
  Calcium: follow- up (Day 6) | -0.039 (0.0506) | -0.033 (0.1074) | -0.090 (0.1158)
  Chloride: Day 2 | 1.0 (1.07) | 0.5 (2.27) | 2.4 (0.92)
  Chloride: follow- up (Day 6) | -1.6 (2.07) | -0.4 (1.60) | 1.6 (2.62)
  Cholesterol: Day 2 | 0.03885 (0.287412) | -0.26871 (0.539200) | -0.18778 (0.233203)
  Cholesterol: follow- up (Day 6) | -0.27519 (0.477560) | -0.38203 (0.701523) | -0.21691 (0.274776)
  Glucose: Day 2 | 0.09019 (0.622942) | 0.05550 (1.760321) | -1.94944 (2.490078)
  Glucose: follow- up (Day 6) | 0.17344 (0.379258) | -0.32606 (0.340109) | -1.87313 (3.549490)
  Magnesium: Day 2 | -0.009 (0.0285) | -0.052 (0.0742) | -0.001 (0.0732)
  Magnesium: follow- up (Day 6) | -0.014 (0.0297) | 0.005 (0.0457) | -0.006 (0.0758)
  Phosphate: Day 2 | 0.003 (0.0509) | 0.080 (0.0953) | 0.105 (0.1872)
  Phosphate: follow- up (Day 6) | -0.005 (0.0682) | -0.064 (0.1421) | -0.106 (0.1897)
  Potassium: Day 2 | -0.11 (0.356) | -0.12 (0.266) | -0.34 (0.487)
  Potassium: follow- up (Day 6) | -0.01 (0.181) | 0.16 (0.396) | -0.38 (0.727)
  Sodium: Day 2 | 0.0 (1.60) | -2.8 (1.39) | -0.1 (2.36)
  Sodium: follow- up (Day 6) | -0.6 (1.77) | -0.9 (1.25) | 1.8 (2.76)
  Triglycerides: Day 2 | -0.15538 (0.940507) | 0.06356 (0.222415) | -0.44776 (1.268752)
  Triglycerides: follow- up (Day 6) | -0.23165 (0.875919) | -0.02260 (0.326110) | -0.40539 (0.781335)
  Urea: Day 2 | -0.021 (0.9152) | 0.531 (0.7122) | 0.765 (0.8025)
  Urea: follow- up (Day 6) | -0.213 (1.0149) | 0.149 (0.5849) | 0.340 (0.2570)
  Urea Nitrogen: Day 2 | 0.0000 (0.89505) | 0.5801 (0.71240) | 0.7586 (0.77366)
  Urea Nitrogen: follow- up (Day 6) | -0.2231 (0.99041) | 0.1785 (0.57247) | 0.3570 (0.26987)

18. Secondary Outcome: Change From Baseline in 12-lead Electrocardiogram (ECG) Parameter: Heart Rate
Description: 12-lead ECG recordings were obtained after the participants have rested for at least 5 minutes in supine position by using an ECG machine that automatically calculates the heart rate. Change from baseline in 12-lead ECG parameter: heart rate at Day 1 and Day 6 were reported.
Time Frame: Baseline, Day 1 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
beats per minute
  Day 1 | 0.3 (5.18) | -0.9 (5.33) | 0.9 (2.70)
  Follow- up (Day 6) | 11.8 (11.02) | 7.4 (11.34) | 5.8 (6.34)

19. Secondary Outcome: Change From Baseline in 12-lead Electrocardiogram (ECG) Parameters: PQ/PR Interval, QRS Duration, QT Interval, Corrected QT Interval Using Fridericia's Formula (QTcF) and RR Duration at Day 1 and Day 6
Description: 12-lead ECG recordings were obtained after the participants have rested for at least 5 minutes in supine position by using an ECG machine that automatically measures PQ/PR, QRS, QT, and QTc intervals and RR duration. Change From Baseline in 12-ECG parameters: PQ/PR interval, QRS duration, QT interval, QTcF interval and RR duration at Day 1 and Day 6 were reported.
Time Frame: Baseline, Day 1 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
milliseconds
  PQ/PR Duration: Day 1 | -0.3 (4.71) | 0.3 (4.46) | -2.0 (17.47)
  PQ/PR Duration: follow-up (Day 6) | -12.5 (11.05) | -4.5 (9.78) | -10.0 (13.52)
  QRS Duration :Day 1 | 0.0 (3.21) | 2.3 (5.06) | 6.5 (9.06)
  QRS Duration: follow-up (Day 6) | -1.3 (3.01) | 3.0 (8.28) | -2.0 (7.63)
  QT Duration: Day 1 | -7.3 (17.33) | -0.3 (11.97) | -0.5 (12.99)
  QT Duration: follow-up (Day 6) | -24.3 (18.77) | -5.5 (22.72) | -7.0 (20.45)
  QTcF - Fridericia's Correction Formula: Day 1 | -6.8 (20.11) | -1.8 (4.89) | 1.5 (11.76)
  QTcF - Fridericia's Correction Formula: follow-up (Day 6) | -2.4 (9.98) | 9.1 (11.49) | 2.9 (15.61)
  RR Duration: Day 1 | -6.1 (79.08) | 9.0 (92.82) | -11.0 (37.85)
  RR Duration: follow-up (Day 6) | -148.1 (126.54) | -87.4 (130.73) | -67.4 (91.17)

20. Secondary Outcome: Change From Baseline in Vital Sign Parameters: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Change from baseline in SBP and DBP at Days 1, 2 and 6 were reported.
Time Frame: Baseline, Day 1, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
millimeters of mercury (mmHg)
  SBP: Day 1 | 3.5 (12.95) | -3.6 (3.58) | 2.0 (6.70)
  SBP: Day 2 | 5.6 (6.97) | 4.8 (13.05) | -1.1 (8.68)
  SBP: follow-up (Day 6) | 0.1 (15.58) | 4.8 (5.99) | 0.9 (13.21)
  DBP: Day 1 | 1.4 (6.86) | -3.5 (7.17) | -2.0 (4.34)
  DBP: Day 2 | 1.9 (4.58) | 0.6 (5.07) | -1.9 (4.52)
  DBP: follow-up (Day 6) | 1.0 (7.37) | 3.3 (4.74) | 0.5 (7.73)

21. Secondary Outcome: Change From Baseline in Vital Sign Parameter: Pulse Rate
Description: Pulse rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Change from baseline in vital sign parameter: pulse rate at Days 1, 2 and 6 were reported.
Time Frame: Baseline, Day 1, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
beats per minute
  Day 1 | 1.1 (2.42) | 1.5 (8.26) | -1.4 (5.53)
  Day 2 | 11.3 (5.18) | 7.4 (7.78) | 8.8 (5.34)
  Follow-up (Day 6) | 11.0 (8.07) | 3.6 (7.31) | 5.9 (6.17)

22. Secondary Outcome: Change From Baseline in Vital Sign Parameter: Respiratory Rate
Description: Respiratory rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Change from baseline in vital sign parameter: respiratory rate at Days 1, 2 and 6 were reported.
Time Frame: Baseline, Day 1, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
breaths per minute
  Day 1 | -1.0 (1.69) | 0.9 (1.64) | -0.6 (1.30)
  Day 2 | 1.5 (2.33) | 0.0 (1.51) | -0.8 (2.43)
  Follow-up (Day 6) | 1.0 (3.02) | -0.5 (0.93) | -0.1 (1.46)

23. Secondary Outcome: Change From Baseline in Vital Sign Parameter: Temperature
Description: Temperature was measured in the semi-supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Change from baseline in vital sign parameter: temperature at Days 1, 2 and 6 were reported.
Time Frame: Baseline, Day 1, Day 2 and follow-up (Day 6)
Population: SAF included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
degree celsius
  Day 1 | -0.04 (0.366) | -0.00 (0.438) | -0.01 (0.270)
  Day 2 | 0.46 (0.463) | 0.05 (0.396) | 0.19 (0.348)
  Follow-up (Day 6) | 0.21 (0.223) | 0.14 (0.444) | 0.16 (0.354)

24. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of M2951
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 32.0 hours post-dose
Population: The PK Population was a subset of the SAF analysis population and consisted of all participants who received at least one dose of active IMP and provide at least one measurable post-dose concentration. A measurement BLQ was considered a valid measurement.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
hours | 2.00 [1.00 to 4.00] | 1.76 [0.500 to 3.02] | 1.75 [1.00 to 3.00]

25. Secondary Outcome: Apparent Elimination Half Life (t1/2) of M2951
Description: T1/2 was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 32.0 hours post-dose
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
hours | 1.54 [1.02 to 1.67] | 2.55 [1.55 to 6.56] | 2.65 [1.81 to 3.02]

26. Secondary Outcome: Area Under The Plasma Concentration-Time Curve From Time Zero to Time 12 Hours (AUC0-12) of M2951
Description: AUC0-12 of M2951 was defined as the area under the plasma concentration time curve from time 0 to 12 hours post-dose.
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0 and 12.0 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 184 (23.6) | 224 (59.7) | 351 (21.7)

27. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time 24 Hours (AUC0-24) of M2951
Description: AUC0-24 of M2951 was defined as the area under the plasma concentration time curve from time 0 to 24 hours post-dose.
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0 and 24.0 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 185 (23.8) | 231 (60.1) | 360 (22.0)

28. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-tlast) of M2951
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-tlast was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 32.0 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 184 (23.9) | 228 (60.9) | 357 (22.3)

29. Secondary Outcome: Apparent Total Body Clearance (CL/f) of M2951
Description: CL/f was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. CL/f was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-t + Clast pred/Lambda Z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the lower limit of quantification (LLOQ) and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 32.0 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
liter per hour (L/h) | 162 (23.6) | 129 (60.6) | 82.9 (21.8)
Statistical Analysis 1: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 2: Mild Hepatic Impairment (Child-Pugh Class A); Mild Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 0.80, 90% CI 2-sided [0.55 to 1.17]
Statistical Analysis 2: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 3: Moderate Hepatic Impairment (Child-Pugh Class B); Moderate Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 0.51, 90% CI 2-sided [0.42 to 0.63]

30. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (VZ/f) of M2951
Description: Vz/f is defined as the distribution of a study drug between plasma and the rest of the body after oral dosing. Vz/f = Dose/(AUC0-infinity multiply by Lambda z) following single dose. AUC0-inf was calculated by combining AUC0-tlast and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 32.0 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
liters | 337 (15.2) | 498 (53.4) | 301 (27.0)

31. Secondary Outcome: Fraction of Unbound Drug (fu) of M2951
Description: fu is defined as the ratio of unbound drug concentration to the total drug concentration.
Time Frame: 1.5, 4, and 12 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of unbound drug
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
ratio of unbound drug | 5.00 (15.3) | 5.78 (17.9) | 6.55 (11.9)

32. Secondary Outcome: Area Under Plasma Concentration for Unbound Drug (M2951) From Time Zero to Infinity (AUC0-inf,u)
Description: AUC0-inf,u was calculated as fu * AUC0-inf. fu was defined as the ratio of unbound drug concentration to the total drug concentration. AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: 1.5, 4, and 12 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 9.28 (30.3) | 13.4 (71.7) | 23.7 (28.5)
Statistical Analysis 1: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 2: Mild Hepatic Impairment (Child-Pugh Class A); Mild Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 1.44, 90% CI 2-sided [0.93 to 2.25]
Statistical Analysis 2: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 3: Moderate Hepatic Impairment (Child-Pugh Class B); Moderate Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 2.55, 90% CI 2-sided [1.98 to 3.29]

33. Secondary Outcome: Maximum Observed Plasma Concentration of Unbound M2951 (Cmax, u)
Description: Cmax,u was calculated as fu * Cmax. fu was defined as the ratio of unbound drug concentration to the total drug concentration. Cmax was obtained directly from the concentration versus time curve.
Time Frame: 1.5, 4, and 12 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 3.19 (22.8) | 4.57 (92.6) | 7.72 (36.1)
Statistical Analysis 1: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 2: Mild Hepatic Impairment (Child-Pugh Class A); Mild Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 1.43, 90% CI 2-sided [0.86 to 2.39]
Statistical Analysis 2: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 3: Moderate Hepatic Impairment (Child-Pugh Class B); Moderate Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 2.42, 90% CI 2-sided [1.87 to 3.14]

34. Secondary Outcome: Apparent Oral Clearance (CL,u/F) of Unbound M2951
Description: CL,u/F was calculated as Dose divided by AUC0-inf, u. AUC0-inf,u was calculated as fu * AUC0-inf. fu was defined as the ratio of unbound drug concentration to the total drug concentration. AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: 1.5, 4, and 12 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 8 | 8 | 8
L/h | 3230 (30.3) | 2240 (71.7) | 1270 (28.5)
Statistical Analysis 1: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 2: Mild Hepatic Impairment (Child-Pugh Class A); Mild Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 0.69, 90% CI 2-sided [0.45 to 1.08]
Statistical Analysis 2: Comparison: Group 1: Normal Hepatic Function (Reference) vs Group 3: Moderate Hepatic Impairment (Child-Pugh Class B); Moderate Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Ratio of geometric least square mean = 0.39, 90% CI 2-sided [0.30 to 0.50]

ADVERSE EVENTS:
Time Frame: up to follow-up (Day 6)
Arm/Group | Group 1: Normal Hepatic Function (Reference) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Normal Hepatic Function (Reference) (N=8) | Group 2: Mild Hepatic Impairment (Child-Pugh Class A) (N=8) | Group 3: Moderate Hepatic Impairment (Child-Pugh Class B) (N=8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Submission of publications to Merck for review at least 60 days prior planned publication. Merck has to provide feedback within 60 days, if any confidential information other than study data is concerned. Should any patent rights be effected, Merck has right to delay publication for another 60 days for patent filing.

DOCUMENTS (2):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04546789/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT04546789/SAP_001.pdf